CLINICAL TRIAL: NCT04113642
Title: The Effect of Activation of Thoracolumbar Fascia on the Thickness of Abdominal Muscles; an Ultrasonographic Study
Brief Title: The Effect Thoracolumbar Fascia on the Abdominal Muscle
Status: Completed | Type: Observational
Sponsor: Koç University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019.100.IRB1.012
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2019-10

CONDITIONS: Abdominal Muscle; Posture; Muscle Strength
Keywords: abdominal muscles; ultrasonography; exercise; lumbar fascia
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- single group: healthy subjects
  Interventions: Other: ultrasonographic measurement of abdominal muscle thickness at four positions

INTERVENTIONS:
Other: ultrasonographic measurement of abdominal muscle thickness at four positions — Thickness of transversus abdominis, internal oblique and external oblique muscles were evaluated using ultrasound at rest and during abdominal hollowing, bridge, and bridge with isometric arm extension.

SUMMARY:
The aim of this study was to evaluate the changes in the thickness of abdominal muscles during activation of thoracolumbar fascia through contracting the gluteus maximus and latissimus dorsi muscles. The hypothesis was that the thickness of transversus abdominis and internal oblique would show greater increase when abdominal contraction was performed with simultaneous contraction of gluteus maximus and latissimus dorsi (bridge with arm extension) than that of abdominal contraction alone (abdominal hollowing) or abdominal contraction with simultaneous activation of only gluteus maximus (bridge). Thirty healthy subjects (15 women, 15 men) were enrolled in this cross-sectional study. Thickness of transversus abdominis, internal oblique and external oblique muscles were evaluated using ultrasound at rest and during three exercise positions: abdominal hollowing in neutral spine, bridge, and bridge with isometric arm extension using ultrasound device equipped with 55 mm convex array transducer

DETAILED DESCRIPTION:
Spinal stabilization is crucial in maintaining healthy posture. Core muscle activation could be enhanced using thoracolumbar fascia for this stability.

Core, also called 'power house', is a muscular box built from abdominal muscles in the front, paraspinal, and gluteal muscles at the back, diaphragm at the top, and pelvic floor muscles at the bottom. Deep core muscles control intersegmental motion and respond to postural and extrinsic load changes and consist of transversus abdominis, internal oblique, multifidi and pelvic floor muscles.

Myofascial system links latissimus dorsi and gluteus maximus through thoracolumbar fascia causing tensegrity-like network in the whole body.

The aim of this study was to evaluate the changes in the thickness of abdominal muscles during activation of thoracolumbar fascia through contracting the gluteus maximus and latissimus dorsi muscles. The hypothesis was that the thickness of transversus abdominis and internal oblique would show greater increase when abdominal contraction was performed with simultaneous contraction of gluteus maximus and latissimus dorsi (bridge with arm extension) than that of abdominal contraction alone (abdominal hollowing) or abdominal contraction with simultaneous activation of only gluteus maximus (bridge).

Thirty healthy subjects (15 women, 15 men) were enrolled in this cross-sectional study. Thickness of transversus abdominis, internal oblique and external oblique muscles were evaluated using ultrasound at rest and during three exercise positions: abdominal hollowing in neutral spine, bridge, and bridge with isometric arm extension using ultrasound device equipped with 55 mm convex array transducer.

ELIGIBILITY:
age of >18 years absence of back or abdominal problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy hospital staff
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Change in ultrasonographic thickness of abdominal muscles | 1 day (Change of muscle thickness from rest to exercise positions)
  The ultrasound transducer was placed over an intersection point of two imaginary lines: one line passing horizontally from the level of navel and the second line running vertically through the anterior superior iliac spine. Subsequent images were obtained at rest, during abdominal hollowing, bridge and bridge with arm extension. Thicknesses of the muscles were measured using onscreen caliper. Results were recorded in millimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Ozden Ozyemisci Taskiran, Prof, Principal Investigator — Koc University School of Medicine
Locations (1):
- Koc University School of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It was not planned to share individual participant data.

REFERENCES:
- [Background] Panjabi MM. Clinical spinal instability and low back pain. J Electromyogr Kinesiol. 2003 Aug;13(4):371-9. doi: 10.1016/s1050-6411(03)00044-0. PMID 12832167
- [Background] Crisco JJ, Panjabi MM, Yamamoto I, Oxland TR. Euler stability of the human ligamentous lumbar spine. Part II: Experiment. Clin Biomech (Bristol). 1992 Feb;7(1):27-32. doi: 10.1016/0268-0033(92)90004-N. PMID 23915613
- [Background] Key J. 'The core': understanding it, and retraining its dysfunction. J Bodyw Mov Ther. 2013 Oct;17(4):541-59. doi: 10.1016/j.jbmt.2013.03.012. Epub 2013 Jun 28. PMID 24139017
- [Background] Akuthota V, Ferreiro A, Moore T, Fredericson M. Core stability exercise principles. Curr Sports Med Rep. 2008 Feb;7(1):39-44. doi: 10.1097/01.CSMR.0000308663.13278.69. PMID 18296944
- [Background] Czaprowski D, Afeltowicz A, Gebicka A, Pawlowska P, Kedra A, Barrios C, Hadala M. Abdominal muscle EMG-activity during bridge exercises on stable and unstable surfaces. Phys Ther Sport. 2014 Aug;15(3):162-8. doi: 10.1016/j.ptsp.2013.09.003. Epub 2013 Sep 27. PMID 24268641
- [Background] Panjabi MM. The stabilizing system of the spine. Part II. Neutral zone and instability hypothesis. J Spinal Disord. 1992 Dec;5(4):390-6; discussion 397. doi: 10.1097/00002517-199212000-00002. PMID 1490035
- [Background] Panjabi M, Abumi K, Duranceau J, Oxland T. Spinal stability and intersegmental muscle forces. A biomechanical model. Spine (Phila Pa 1976). 1989 Feb;14(2):194-200. doi: 10.1097/00007632-198902000-00008. PMID 2922640
- [Background] Schleip R, Muller DG. Training principles for fascial connective tissues: scientific foundation and suggested practical applications. J Bodyw Mov Ther. 2013 Jan;17(1):103-15. doi: 10.1016/j.jbmt.2012.06.007. Epub 2012 Jul 21. PMID 23294691
- [Background] Dischiavi SL, Wright AA, Hegedus EJ, Bleakley CM. Biotensegrity and myofascial chains: A global approach to an integrated kinetic chain. Med Hypotheses. 2018 Jan;110:90-96. doi: 10.1016/j.mehy.2017.11.008. Epub 2017 Nov 20. PMID 29317079
- [Background] Bogduk N, Macintosh JE. The applied anatomy of the thoracolumbar fascia. Spine (Phila Pa 1976). 1984 Mar;9(2):164-70. doi: 10.1097/00007632-198403000-00006. PMID 6729580
- [Background] Wilke J, Krause F, Vogt L, Banzer W. What Is Evidence-Based About Myofascial Chains: A Systematic Review. Arch Phys Med Rehabil. 2016 Mar;97(3):454-61. doi: 10.1016/j.apmr.2015.07.023. Epub 2015 Aug 14. PMID 26281953
- [Background] Escamilla RF, Lewis C, Bell D, Bramblet G, Daffron J, Lambert S, Pecson A, Imamura R, Paulos L, Andrews JR. Core muscle activation during Swiss ball and traditional abdominal exercises. J Orthop Sports Phys Ther. 2010 May;40(5):265-76. doi: 10.2519/jospt.2010.3073. PMID 20436242
- [Background] Hodges PW, Pengel LH, Herbert RD, Gandevia SC. Measurement of muscle contraction with ultrasound imaging. Muscle Nerve. 2003 Jun;27(6):682-92. doi: 10.1002/mus.10375. PMID 12766979
- [Background] Ferreira PH, Ferreira ML, Nascimento DP, Pinto RZ, Franco MR, Hodges PW. Discriminative and reliability analyses of ultrasound measurement of abdominal muscles recruitment. Man Ther. 2011 Oct;16(5):463-9. doi: 10.1016/j.math.2011.02.010. Epub 2011 Mar 12. PMID 21398167
- [Background] Chanthapetch P, Kanlayanaphotporn R, Gaogasigam C, Chiradejnant A. Abdominal muscle activity during abdominal hollowing in four starting positions. Man Ther. 2009 Dec;14(6):642-6. doi: 10.1016/j.math.2008.12.009. Epub 2009 Feb 28. PMID 19251466
- [Background] Hodges PW. Ultrasound imaging in rehabilitation: just a fad? J Orthop Sports Phys Ther. 2005 Jun;35(6):333-7. doi: 10.2519/jospt.2005.0106. No abstract available. PMID 16001904
- [Background] Costa LO, Maher CG, Latimer J, Smeets RJ. Reproducibility of rehabilitative ultrasound imaging for the measurement of abdominal muscle activity: a systematic review. Phys Ther. 2009 Aug;89(8):756-69. doi: 10.2522/ptj.20080331. Epub 2009 Jun 11. PMID 19520732
- [Background] Linek P, Saulicz E, Wolny T, Mysliwiec A. Intra-rater reliability of B-mode ultrasound imaging of the abdominal muscles in healthy adolescents during the active straight leg raise test. PM R. 2015 Jan;7(1):53-9. doi: 10.1016/j.pmrj.2014.07.007. Epub 2014 Aug 1. PMID 25088316
- [Background] Linek P, Saulicz E, Wolny T, Mysliwiec A. Reliability of B-mode sonography of the abdominal muscles in healthy adolescents in different body positions. J Ultrasound Med. 2014 Jun;33(6):1049-56. doi: 10.7863/ultra.33.6.1049. PMID 24866612
- [Background] Gibbon KC, Debuse D, Hibbs A, Caplan N. Reliability and Precision of Sonography of the Lumbar Multifidus and Transversus Abdominis During Dynamic Activities. J Ultrasound Med. 2017 Mar;36(3):571-581. doi: 10.7863/ultra.16.03059. Epub 2017 Feb 2. PMID 28150321
- [Background] Mangum LC, Sutherlin MA, Saliba SA, Hart JM. Reliability of Ultrasound Imaging Measures of Transverse Abdominis and Lumbar Multifidus in Various Positions. PM R. 2016 Apr;8(4):340-347. doi: 10.1016/j.pmrj.2015.09.015. Epub 2015 Sep 30. PMID 26428485
- [Background] Kim JS, Seok CH, Jeon HS. Abdominal draw-in maneuver combined with simulated weight bearing increases transversus abdominis and internal oblique thickness. Physiother Theory Pract. 2017 Dec;33(12):954-958. doi: 10.1080/09593985.2017.1359866. Epub 2017 Sep 6. PMID 28876160
- [Background] Gnat R, Saulicz E, Miadowicz B. Reliability of real-time ultrasound measurement of transversus abdominis thickness in healthy trained subjects. Eur Spine J. 2012 Aug;21(8):1508-15. doi: 10.1007/s00586-012-2184-4. Epub 2012 Feb 12. PMID 22327252
- [Background] O'Sullivan PB. Lumbar segmental 'instability': clinical presentation and specific stabilizing exercise management. Man Ther. 2000 Feb;5(1):2-12. doi: 10.1054/math.1999.0213. PMID 10688954
- [Background] Teyhen DS, Miltenberger CE, Deiters HM, Del Toro YM, Pulliam JN, Childs JD, Boyles RE, Flynn TW. The use of ultrasound imaging of the abdominal drawing-in maneuver in subjects with low back pain. J Orthop Sports Phys Ther. 2005 Jun;35(6):346-55. doi: 10.2519/jospt.2005.35.6.346. PMID 16001906
- [Background] Panjabi MM. The stabilizing system of the spine. Part I. Function, dysfunction, adaptation, and enhancement. J Spinal Disord. 1992 Dec;5(4):383-9; discussion 397. doi: 10.1097/00002517-199212000-00001. PMID 1490034
- [Background] Barker PJ, Briggs CA, Bogeski G. Tensile transmission across the lumbar fasciae in unembalmed cadavers: effects of tension to various muscular attachments. Spine (Phila Pa 1976). 2004 Jan 15;29(2):129-38. doi: 10.1097/01.BRS.0000107005.62513.32. PMID 14722403
- [Background] Vleeming A, Pool-Goudzwaard AL, Stoeckart R, van Wingerden JP, Snijders CJ. The posterior layer of the thoracolumbar fascia. Its function in load transfer from spine to legs. Spine (Phila Pa 1976). 1995 Apr 1;20(7):753-8. PMID 7701385
- [Background] Barker PJ, Hapuarachchi KS, Ross JA, Sambaiew E, Ranger TA, Briggs CA. Anatomy and biomechanics of gluteus maximus and the thoracolumbar fascia at the sacroiliac joint. Clin Anat. 2014 Mar;27(2):234-40. doi: 10.1002/ca.22233. Epub 2013 Aug 20. PMID 23959791
- [Background] Stecco A, Gilliar W, Hill R, Fullerton B, Stecco C. The anatomical and functional relation between gluteus maximus and fascia lata. J Bodyw Mov Ther. 2013 Oct;17(4):512-7. doi: 10.1016/j.jbmt.2013.04.004. Epub 2013 May 11. PMID 24139012
- [Background] Bogduk N, Johnson G, Spalding D. The morphology and biomechanics of latissimus dorsi. Clin Biomech (Bristol). 1998 Sep;13(6):377-385. doi: 10.1016/s0268-0033(98)00102-8. PMID 11415812
- [Background] Carvalhais VO, Ocarino Jde M, Araujo VL, Souza TR, Silva PL, Fonseca ST. Myofascial force transmission between the latissimus dorsi and gluteus maximus muscles: an in vivo experiment. J Biomech. 2013 Mar 15;46(5):1003-7. doi: 10.1016/j.jbiomech.2012.11.044. Epub 2013 Feb 8. PMID 23394717